CLINICAL TRIAL: NCT00268359
Title: Bevacizumab in Combination With Irinotecan for Malignant Gliomas
Brief Title: Bevacizumab and Irinotecan in Treating Patients With Recurrent or Refractory Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: Pro00004091; DUMC-6771-05-1R0; GENENTECH-AVF3311s; CDR0000450832 (Other: NCI)
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2013-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult glioblastoma; adult gliosarcoma; recurrent adult brain tumor; adult giant cell glioblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Bevacizumab; Irinotecan

INTERVENTIONS:
Biological: bevacizumab
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Drugs used in chemotherapy, such as irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bevacizumab together with irinotecan may kill more tumors cells.

PURPOSE: This phase II trial is studying the side effects of bevacizumab and how well giving bevacizumab together with irinotecan works in treating patients with recurrent or refractory gliomas.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of bevacizumab and irinotecan hydrochloride in patients with recurrent or refractory grade 3 or 4 malignant gliomas.

Secondary

* Determine the activity of this regimen, in terms of progression-free survival, in these patients.

OUTLINE: Patients receive bevacizumab and irinotecan hydrochloride every 2 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 68 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary grade 3 or 4 malignant glioma of 1 of the following types:

  * Glioblastoma multiforme
  * Gliosarcoma
  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
* Patients with recurrent disease whose original diagnostic pathology confirmed malignant glioma will not need re-biopsy
* Measurable recurrent or residual primary disease on contrast-enhanced MRI or CT scan
* Failed ≥ 1 prior chemotherapy regimen (with or without radiotherapy)

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Hematocrit > 29%
* Absolute neutrophil count > 1,500/mm^3
* Platelets > 125,000/mm^3
* Serum SGOT and bilirubin < 1.5 times upper limit of normal
* Creatinine < 1.5 mg/dL
* Urine protein:creatinine ratio ≤ 1.0
* Blood pressure ≤ 150/100 mmHg
* No unstable angina
* No New York Heart Association class II or greater congestive heart failure
* No myocardial infarction within the past 6 months
* No stroke within the past 6 months
* No clinically significant peripheral vascular disease
* No evidence of bleeding diathesis or coagulopathy
* No significant traumatic injury within the past 28 days

PRIOR CONCURRENT THERAPY:

* At least 4 weeks must have elapsed since prior chemotherapy or radiotherapy unless there is unequivocal evidence of tumor progression
* At least 6 weeks since prior surgical resection
* No previous major surgical procedures or open biopsies within 28 days prior to study entry
* No previous minor surgical procedures, fine needle aspirations, or core biopsies within 7 days prior to study entry
* No anticipated need for major surgical procedures during the course of the study
* No concurrent aspirin, non-steroidal anti-inflammatory drugs, or clopidogrel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2005-05; Primary Completion 2006-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Safety
Activity in terms of progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: James J. Vredenburgh, MD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Desjardins A, Reardon DA, Herndon JE 2nd, Marcello J, Quinn JA, Rich JN, Sathornsumetee S, Gururangan S, Sampson J, Bailey L, Bigner DD, Friedman AH, Friedman HS, Vredenburgh JJ. Bevacizumab plus irinotecan in recurrent WHO grade 3 malignant gliomas. Clin Cancer Res. 2008 Nov 1;14(21):7068-73. doi: 10.1158/1078-0432.CCR-08-0260. PMID 18981004
- [Result] Sathornsumetee S, Cao Y, Marcello JE, Herndon JE 2nd, McLendon RE, Desjardins A, Friedman HS, Dewhirst MW, Vredenburgh JJ, Rich JN. Tumor angiogenic and hypoxic profiles predict radiographic response and survival in malignant astrocytoma patients treated with bevacizumab and irinotecan. J Clin Oncol. 2008 Jan 10;26(2):271-8. doi: 10.1200/JCO.2007.13.3652. PMID 18182667
- [Result] Vredenburgh JJ, Desjardins A, Herndon JE 2nd, Dowell JM, Reardon DA, Quinn JA, Rich JN, Sathornsumetee S, Gururangan S, Wagner M, Bigner DD, Friedman AH, Friedman HS. Phase II trial of bevacizumab and irinotecan in recurrent malignant glioma. Clin Cancer Res. 2007 Feb 15;13(4):1253-9. doi: 10.1158/1078-0432.CCR-06-2309. PMID 17317837